CLINICAL TRIAL: NCT02205697
Title: Theory of Planned Behavior and Implementation Intentions: Effective for Improving Fruit and Vegetable Intake in Women of Low Socioeconomic Status?
Brief Title: Theory of Planned Behavior and Implementation Intentions
Acronym: TPBIIFV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: mdh-32828
Record Dates: First submitted 2014-07-29; First posted 2014-07-31 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2015-07

CONDITIONS: Dietary Modification
Keywords: Fruit; Vegetable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Implementation intention (Experimental): The entire cohort will be asked to create an implementation intention to increase their intake of fruit and vegetables over the study period.
  Interventions: Behavioral: Implementation intention

INTERVENTIONS:
Behavioral: Implementation intention — The intervention consists of an implementation intention whereby subjects create a unique plan to increase their fruit and vegetable intake by planning the where, when, and what to increase their fruit and vegetable intake.

SUMMARY:
Diet quality has been associated with a variety of chronic diseases including obesity. One measure that has been studied as an indicator for diet quality is fruit and vegetable intake. Although the US government has suggested that American's increase their intake of fruit and vegetables, epidemiological data suggest that most Americans have not been successful doing do, with the strongest disparity seen in people of low socioeconomic status (SES). This disparity in fruit and vegetable intake is thought to be the result of both individual and environmental factors that influence this health behavior. To help decrease the disparate rise in incidence of chronic disease in people of low SES, effective, cost-efficient and easy to implement interventions to improve fruit and vegetable intake and diet quality are needed.

Theoretical models of health behavior change have been successfully used in research targeting individual factors associated with health behaviors. One theory, the Theory of Planned Behavior (TPB), and a proposed extension of this model (implementation intentions) have been shown to be effective to increase fruit and vegetable intake in (mostly) white adults of average socioeconomic status. It is not know whether an implementation intention intervention to increase fruit and vegetable intake would be effective in women who are of low socioeconomic status. The primary aim of this research is to study (using quantitative and qualitative analysis) an implementation intention intervention to produce a positive change in fruit and vegetable intake. We theorize that the setting of an implementation intention in this group will be effective, cost-effective, and easy to implement intervention to promote an increase in fruit and vegetable intake.

DETAILED DESCRIPTION:
Theory of Planned Behavior Variables (attitude, perceived behavioral control, intention) measured via survey using 1 question each, bivariate semantic differential scale.

Main outcomes measure is fruit and vegetable intake. Behavioral Risk Factor Surveillance System Fruit and Vegetable Module (6-item screener) + pictorial of serving sizes.

Demographic data measured via survey. Height measured via tape measure. Weight measured using a standing scale.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Boston Public Housing
* Identifies as female
* Age 18-72
* Able to give informed consent
* Agrees to be randomized into either the intervention or the control groups
* Understands English sufficient to comprehend purpose, risks, benefits and voluntary nature of the study, and to complete the surveys and provide information in this language

Exclusion Criteria:

* Does not consent to study participation
* Currently pregnant
* Identifies as following a strict medically prescribed diet, as having an allergy to fruit and/or vegetables, or as currently taking medications that necessitate the avoidance or reduction of fruit and/or vegetable intake.
* Does not agree to be randomized into either the intervention or control groups

Ages: 18 Years to 72 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in mean intake of fruit and vegetables (servings per day) both within and between the experimental and control groups. | 30 days
  Change in mean intake of fruit and vegetables (servings per day) will be assessed in both the experimental and control groups using the Behavioral Risk Factor Surveillance System (BRFSS) Fruit and Vegetable Module. Inferential statistics will be used to assess differences in change in mean fruit and vegetable intake both within and between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Michele A DeBiasse, MS, RDN, Principal Investigator — Boston University/Graduate Medical Sciences
Locations (1):
- Boston University School of Medicine, Boston, Massachusetts, United States